CLINICAL TRIAL: NCT03468699
Title: Outcomes of Autologous Bone Marrow Mononuclear Stem Cell (BMMC) Transplantation for Children Suffering From Liver Cirrhosis Due to Biliary Atresia After Kasai's Operation: An Open Label Uncontrolled Clinical Trial
Brief Title: Autologous Bone Marrow Mononuclear Stem Cell for Children Suffering From Liver Cirrhosis Due to Biliary Atresia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VinmecRISCGT78
Record Dates: First submitted 2018-01-26; First posted 2018-03-16 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Liver Cirrhosis, Biliary
Keywords: Autologous bone marrow Transplantation; biliary atresia; Kasai's operation; liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Biliary Atresia; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous BMMC transplantation (Experimental): Stem cell transplantations include 2 administrations of autologous bone marrow mononuclear cells via the hepatic artery at baseline and 6 months afterward
  Interventions: Combination Product: Autologous BMMC transplantation

INTERVENTIONS:
Combination Product: Autologous BMMC transplantation — Stem cell transplantation

SUMMARY:
The aim of this study was to evaluate the safety and effectiveness of autologous bone marrow mononuclear stem cell transplantation for Children Suffering from Liver Cirrhosis Due to Biliary Atresia

DETAILED DESCRIPTION:
This study is ferformed to evaluate the safety and effectiveness of autologous bone marrow mononuclear stem cell transplantation in the management of Liver Cirrhosis Due to Biliary Atresia after Kasai's operation of 20 patients at Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Vietnam from January 2017 to December 2018

ELIGIBILITY:
Inclusion Criteria:

* Children were diagnosed with Liver Cirrhosis Due to biliary atresia after Kasai's operation
* From 5 months to 2 years old
* Weight ≥ 6 kg
* Patients with manifestation of cirrhosis after Kasai's operation: hepatomegaly, congestive splenomegaly, elevated liver enzymes, Esophageal Varices (based on Endoscopic Diagnosis), cirrhosis (based on liver biopsy)

Exclusion Criteria:

* Under 1 year old patients
* Epilepsy
* Coagulation disorders
* Allergy to anesthetic agents
* Severe health conditions such as cancer, failure of heart, lung, liver or kidney
* Active infections
* Severe psychiatric disorders

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Assess the changes in cholestasis | Baseline, 3, 6 months and 12 months after transplantation
  Using Bilirubin (total, direct and indirect) (units: mg/dL) to measure the changes in cholestasis
Assess the changes in Liver function | Baseline, 3, 6 months and 12 months after transplantation
  Using AST (Aspart transaminase) and ALT (Alanin transaminase) (units: U/L), GGT (Gamma GT) (units: UI/L), and Bilirubin (units: mg/dL) to measure the changes in Liver function
Assess the changes in level of cirrhosis | Baseline, 3, 6 months and 12 months after transplantation
  Using PELD score (according to the suggestion of The Liver and Intestinal Organ Transplantation Committee in 2009). PELD is calculated based on three indicators: albumin (g / dL), bilirubin (units: mg / dL) and INR (international normalized ratio). Formula: PELD = 10 * (0.48 * ln(Serum Bilirubin) + 1.857 * ln(INR) - 0.687 * ln(Albumin) + (0.436 if patient is less than 1 year old) + (0.667 if patient has growth failure)). Evaluate the result:
  * If PELD <10: good results
  * If 10 <PELD <15: average results
  * If PELD> 15: bad results
  Albumin (Unit: g / dL), bilirubin (units: mg / dL) and INR (international normalized ratio).
Assess the changes in liver biopsy | Baseline, 3, 6 months and 12 months after transplantation
  Liver biopsy, in combination with history and physical examination data, is a powerful clinical tool for diagnosing and treating liver disease to evaluate the changes in liver biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Liem Nguyen, Principal Investigator — Vinmec Research Institute of Stem Cell and Gene Technology
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Vietnam

REFERENCES:
- [Background] Nicolas C, Wang Y, Luebke-Wheeler J, Nyberg SL. Stem Cell Therapies for Treatment of Liver Disease. Biomedicines. 2016 Jan 6;4(1):2. doi: 10.3390/biomedicines4010002. PMID 28536370
- [Background] Levicar N, Dimarakis I, Flores C, Tracey J, Gordon MY, Habib NA. Stem cells as a treatment for chronic liver disease and diabetes. Handb Exp Pharmacol. 2007;(180):243-62. doi: 10.1007/978-3-540-68976-8_11. PMID 17554512
- [Background] Irfan A, Ahmed I. Could Stem Cell Therapy be the Cure in Liver Cirrhosis? J Clin Exp Hepatol. 2015 Jun;5(2):142-6. doi: 10.1016/j.jceh.2014.03.042. Epub 2014 Mar 27. PMID 26155042
- [Background] Sharma S, Kumar L, Mohanty S, Kumar R, Datta Gupta S, Gupta DK. Bone marrow mononuclear stem cell infusion improves biochemical parameters and scintigraphy in infants with biliary atresia. Pediatr Surg Int. 2011 Jan;27(1):81-9. doi: 10.1007/s00383-010-2712-4. PMID 20857300
- [Background] Khan AA, Parveen N, Mahaboob VS, Rajendraprasad A, Ravindraprakash HR, Venkateswarlu J, Rao P, Pande G, Narusu ML, Khaja MN, Pramila R, Habeeb A, Habibullah CM. Management of hyperbilirubinemia in biliary atresia by hepatic progenitor cell transplantation through hepatic artery: a case report. Transplant Proc. 2008 May;40(4):1153-5. doi: 10.1016/j.transproceed.2008.03.110. PMID 18555137
- [Derived] Nguyen TL, Nguyen HP, Ngo DM, Ha THT, Mai KA, Bui TH, Nguyen PV, Pham LH, Hoang DM, Cao ADT. Autologous bone marrow mononuclear cell infusion for liver cirrhosis after the Kasai operation in children with biliary atresia. Stem Cell Res Ther. 2022 Mar 14;13(1):108. doi: 10.1186/s13287-022-02762-x. PMID 35287722